CLINICAL TRIAL: NCT03442504
Title: Evaluation Study of the Prediction of the Response to Second-line Hormone Therapy by 16α- [18F] Fluoro-17β-estradiol (FES) PET in Patients With Metastatic Breast Cancer
Brief Title: Prediction of Response to 2nd-line Hormone Therapy by FES CT/PET in Patients With Metastatic Breast Cancer
Acronym: TEP-FES
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ICO-N-2016-02
Record Dates: First submitted 2018-02-16; First posted 2018-02-22 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Metastatic Breast Cancer
Keywords: metastatic Breast cancer; FES PET/CT; menopausal patients; recurrence after a 1st line of hormone therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FES PET/CT (Other): The images will be made immediately after the injection of the FES in a dynamic acquisition, of 30 minutes, centered on a positive FDG lesion. The imaging will then be completed 1 hour after the injection, after obtaining a urination, by an acquisition "whole body" (from the top of the skull to the root of the thighs or more if element on FDG or conventional imaging) which will be performed in the supine position with arms around the body. During the PET / CT scan, patients will breathe spontaneously. The acquisition will last 30 minutes.
  Interventions: Diagnostic Test: FES PET/CT

INTERVENTIONS:
Diagnostic Test: FES PET/CT — There will be no premedication or other treatment before and after PET FES. PET / CT will be performed at the center level on a hybrid PET camera.
  * The first TEP FES acquisition begins at the time of injection and continues for 30 minutes,
  * The second acquisition of 20 minutes takes place 60 minutes after the injection is a total of 50 minutes of imaging and 1:30 in the service.

SUMMARY:
Clinicians are currently proposing second-line hormonal treatment to a metastatic patient who is progressing after first-line hormonal therapy if the initial disease was RH + with an increase in survival without recurrence more or less long. The biopsy of the metastatic site or sites is rarely performed because of the heaviness of the gesture. Clinicians are waiting for imaging, which can replace biopsy before the second-line metastatic hormone treatment in breast cancer, which will reveal the metastatic lesion heterogeneity allowing to establish if hormone therapy is the best therapeutic option for these patients and therefore lead to a personalized medicine driven by PET FES. This imaging approach seems all the more interesting as ER expression appears to evolve over time under the pressure of treatment or the natural evolution of carcinomas.

Currently, no studies in breast cancer, in an ER + population on the initial tumor and Her2 negative, are listed for the study of ER expression by PET FES before a second metastatic hormone treatment line.

DETAILED DESCRIPTION:
Approximately 70% of breast cancer patients have estrogen-receptor-expressing tumors, making hormone therapy an attractive option for adjuvant and metastatic treatment. The expression of estrogen receptors is modified during the course of treatment. Tumor development, there is a discrepancy between primary tumors and metastases from 14.5% to 40% of cases. Biopsies are useful for reassessing a patient's "estrogen receptor" status, but it is not always feasible especially at the stage of multiple metastases and the gesture remains invasive.

The sensitivity and specificity of PET FES has been studied in patients with "estrogen-positive receptor" breast cancer lesions. Sensitivity was good except for liver metastases due to physiological binding of this tracer to the liver. Quantification of FES binding was correlated with expression of estrogen receptors visualized in IHC. Metastases could be seen with FES in the bone, lung and lymph nodes and more difficult in the liver.

Clinicians are currently proposing second-line hormonal treatment to a metastatic patient who is progressing after first-line hormonal therapy if the initial disease was RH + with an increase in survival without recurrence more or less long. The biopsy of the metastatic site or sites is rarely performed because of the heaviness of the gesture. Clinicians are waiting for imaging, which can replace biopsy before the second-line metastatic hormone treatment in breast cancer, which will reveal the metastatic lesion heterogeneity allowing to establish if hormone therapy is the best therapeutic option for these patients and therefore lead to a personalized medicine driven by PET FES. This imaging approach seems all the more interesting as ER expression appears to evolve over time under the pressure of treatment or the natural evolution of carcinomas.

Currently, no studies in breast cancer, in an ER + population on the initial tumor and Her2 negative, are listed for the study of ER expression by PET FES before a second metastatic hormone treatment line.

ELIGIBILITY:
Inclusion Criteria:

1. Primary breast tumor (ductal or lobular) expressing immunohistochemistry of hormone receptors (RP + and / or RE +, with significance level ≥ 10%) but not overexpressing HER2,
2. Metastatic stage with at least one lesion identifiable on the conventional balance sheet other than a liver injury,
3. Patient progressing under a 1st line of hormone therapy,
4. Patient candidate for a new second-line hormonal treatment,
5. Postmenopausal patient,
6. Karnofsky ≥ 70 or ECOG 0-1
7. Life expectancy of at least 6 months
8. Creatinine <= 2.5 normal
9. Social insured patient
10. Signed informed consent

Exclusion Criteria:

1. HER2 overexpressing primary tumor in immunohistochemistry,
2. Tumor that does not significantly (<10%) express the hormonal receptors,
3. Hormonal treatment in progress,
4. Contraindication to a new second-line hormonal treatment,
5. Patient receiving or likely to receive second-line chemotherapy in the course of the evolution of her breast cancer,
6. Persons deprived of liberty or guardianship,
7. Impossibility of submitting to the medical examination of the test for geographical, social or psychological reasons,
8. Serious illness or comorbidity assessed at risk,
9. History of cancer within 5 years, with the exception of cutaneous carcinomas other than melanomas, or carcinoma in situ of the cervix,
10. Intellectual inability to sign informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Determine the predictive value of PET at the "lesion" level | 6 weeks
  Determine the predictive value of PET at the "lesion" level, before a second-line hormonal treatment on the response obtained at 6 weeks of treatment.

SECONDARY OUTCOMES:
Determine the predictive value of PET at FES at the "patient" level | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Caroline ROUSSEAU, MD, Principal Investigator — Institut de Cancérologie de l'Ouest
Locations (4):
- France (4):
  - Institut de Cancerologie de l'Ouest, Angers
  - CHU de Brest, Brest
  - Centre Georges François Leclerc, Dijon
  - ICO René Gauducheau, Saint-Herblain